CLINICAL TRIAL: NCT05807607
Title: Peripheral Nerve and Spinal Cord Stimulation in Patients With Pain Syndrome as a Result of Lower Limb Amputation in Order to Relieve Pain Syndrome and Develop Phantom Pain Biomarkers
Brief Title: Study of Lower-limb Phantom Pain Syndrome Using Peripheral Nerve and Spinal Cord Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Artur Biktimirov (Other)
Responsible Party: Sponsor-Investigator, Artur Biktimirov, Far Eastern Federal University, Far Eastern Federal University
Organization: Far Eastern Federal University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DVFU-10
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Phantom Limb Pain; Phantom Pain; Amputation; Lower Limb Amputation
Keywords: Neurostimulation; Spinal cord stimulation; Peripheral nerve stimulation; Phantom limb pain; Pain suppression; Lower-limb amputation
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who underwent the lower limb amputation and have phantom pain syndrome (Experimental)
  Interventions: Procedure: Implantation of PNS electrodes during surgery, mapping to select sites with the best effect and daily modulation.; Procedure: SCS electrode implantation at surgery, mapping to select sites with the best effect and pain modulation; Procedure: Change according to the scale of the PainDetect questionnaire

INTERVENTIONS:
Procedure: Implantation of PNS electrodes during surgery, mapping to select sites with the best effect and daily modulation. — PNS electrodes are implanted in the area of peripheral nerves of the amputated limb. During phantom pain mapping, multichannel electrodes are used to stimulate peripheral nerves at different sites in the stump. Stimulation turns on sequentially at different stimulation sites; sites are selected where pain is most effectively suppressed. These sites are assigned to the patient for daily modulation.
Procedure: SCS electrode implantation at surgery, mapping to select sites with the best effect and pain modulation — SСS electrodes are implanted in the area of targeted peripheral nerves in the amputated limb. During phantom pain mapping, multichannel electrodes are used to stimulate the spinal cord at different sites. Stimulation starts at a specific site at a frequency of 1 Hz and increases by 0.1 Hz until the patient no longer feels phantom pain. Stimulation turns on sequentially at different stimulation sites; sites are selected where pain is most effectively suppressed. These sites are assigned to the patient for daily modulation.
Procedure: Change according to the scale of the PainDetect questionnaire — This procedure uses the method of electroencephalography (EEG). EEG signals are recorded during the entire experiment. First, the patient is recorded at rest with stimulator on (PNS/SCS) with eyes open and then closed, in the stimulator off state (eyes open, then closed) in order to return the patient to the preoperative state. The stimulation is then turned back on to the original level of pain suppression. The moments of pain suppression are fixed by marking.

SUMMARY:
Brief Summary: The purpose of this study is to evaluate the effectiveness of neuromodulation for relief of phantom limb pain (PLP) using peripheral nerve (PNS) and spinal cord (SCS) stimulation with implantable electrodes. The researchers expect that PLP in patients with lower limb amputation will be relieved by peripheral nerve and the spinal cord stimulation. The possibility of finding EEG biomarkers for phantom pain will be explored.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of neuromodulation for relief of phantom limb pain (PLP) using peripheral nerve (PNS) and spinal cord stimulation (SCS) with implantable electrodes.

The study is conducted to collect information on the role of non-adaptive neuroplasticity and inhibitory descending antinociceptive influences, which determine the effect of peripheral nerve and spinal cord stimulation with implanted electrodes in patients with phantom limb pain as a result of amputation of the lower limb. Neuromodulation is a potential treatment option for chronic pain that may alter maladaptive neuroplasticity and enhance descending inhibitory pathways.

Study participants will be selected according to the inclusion criteria. Next, multichannel electrodes will be implanted in the region of the target peripheral nerves of the amputated limb and the corresponding segments of the spinal cord. The evaluation of the therapeutic effects of pain syndromes will be carried out in the mode of long-term repetitive nerve stimulation. Postoperative follow-up will be carried out from 2 weeks to 1 month. During the follow-up period, patients will complete scales and questionnaires daily.

The stimulator is turned on the day after surgery to assess pain relief. The patient is explained the rules for using the stimulator. The selection of stimulation parameters is carried out according to the generally accepted methodology (the stimulation zone should overlap the pain zone; stimulation should be in the nature of pleasant vibrations). The patient will be given a test stimulation diary to complete every day (at the end of the day) during the entire stimulation period.

The researchers expect that phantom limb pain in patients undergoing lower limb amputation will be relieved by peripheral nerve stimulation. We will explore the possibility of creating a personal phantom sensitivity map to optimize the stimulation program. We will study improving the quality of life and reducing pain.

Patients will be asked to participate in an experiment using electroencephalography (EEG) starting on the 3rd day after implantation. The purpose of this entry is to investigate the biomarkers of phantom pain. As part of the experimental procedure, we plan to sequentially turn off the stimulator until the patient returns to the preoperative pain state, and also turn on the stimulator with fixation of the moments of pain suppression to the level at the beginning of the experiment. During the entire period, the patient's EEG will be recorded. The researchers expect to see changes in alpha and theta EEG rhythms under these experimental conditions.

ELIGIBILITY:
Inclusion criteria for the study:

* Patients with implanted neuromodulation devices.
* Amputation of the lower limb.
* Age ranges from 18 to 65 years old.
* The duration from the moment of amputation is from 12 months.
* The presence of persistent chronic pain syndrome is from 4 to 10 points according to the Visual Analogue Scale
* Absence of pregnancy at the time of implantation, confirmed by a pregnancy test.

Exclusion criteria:

* The presence of severe somatic pathology that prevents surgical treatment and participation in the study.
* The presence of mental illness (including history), severe depression, suicidal tendencies, history of suicide.
* The presence of gross orthopedic deformity in the limb above the amputation level.
* History of oncology.
* History of epilepsy.
* Complicated TBI or history of stroke.
* The impossibility of conducting electrical stimulation due to another somatic pathology.
* Purulent septic pathology.
* Drug addiction (including history).
* Congenital malformation of the lower limb.
* Anomalies in the development of the CNS.
* Any conditions that fall under the exclusion criteria according to the researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Determining the effectiveness of phantom pain suppression based on the Test Stimulation Diary | up to 1 month
  The patient completes a Test Stimulation Diary at the end of each day, noting the location of phantom pain and the percentage of pain reduction during stimulation.
Change according to the scale of the DN4 Neuropathic Pain Questionnaire | : baseline and up to 1 month
  The DN4 Neuropathic Pain Questionnaire defines the neuropathic nature of pain with a point of 4 to 10.
Change according to the scale of the PainDetect questionnaire | up to 1 month
  The PainDetect questionnaire reflects all possible parameters of pain and allows us to very clearly track the picture of the pain syndrome in dynamics. The score is made in the range from 0 (best score) to 38 (worst score) points.
Change in relative power in slow frequencies (alpha and theta ranges) on the EEG with the neurostimulator on/off and eyes open/closed. | up to 1 month
  Data analysis is done in MNE Python. An average reference is used. Artifact correction is carried out using the analysis of independent components. Additionally, band-pass filtering is applied in the range from 1 to 40 Hz. The general analysis pipeline includes the calculation of the normalized power spectral density, after which the average power of the alpha rhythm is divided by the average power of the theta rhythm. This ratio is compared under different experimental conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Federal University (FEFU), Vladivostok, Primorskiy (Maritime) Kray, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Our institution discovers this possibilities to share the data after the study

REFERENCES:
- [Background] Knotkova H, Hamani C, Sivanesan E, Le Beuffe MFE, Moon JY, Cohen SP, Huntoon MA. Neuromodulation for chronic pain. Lancet. 2021 May 29;397(10289):2111-2124. doi: 10.1016/S0140-6736(21)00794-7. PMID 34062145
- [Background] Graczyk EL, Schiefer MA, Saal HP, Delhaye BP, Bensmaia SJ, Tyler DJ. The neural basis of perceived intensity in natural and artificial touch. Sci Transl Med. 2016 Oct 26;8(362):362ra142. doi: 10.1126/scitranslmed.aaf5187. PMID 27797958
- [Background] Mekhail N, Levy RM, Deer TR, Kapural L, Li S, Amirdelfan K, Hunter CW, Rosen SM, Costandi SJ, Falowski SM, Burgher AH, Pope JE, Gilmore CA, Qureshi FA, Staats PS, Scowcroft J, Carlson J, Kim CK, Yang MI, Stauss T, Poree L; Evoke Study Group. Long-term safety and efficacy of closed-loop spinal cord stimulation to treat chronic back and leg pain (Evoke): a double-blind, randomised, controlled trial. Lancet Neurol. 2020 Feb;19(2):123-134. doi: 10.1016/S1474-4422(19)30414-4. Epub 2019 Dec 20. PMID 31870766
- [Background] Ortiz-Catalan M, Mastinu E, Sassu P, Aszmann O, Branemark R. Self-Contained Neuromusculoskeletal Arm Prostheses. N Engl J Med. 2020 Apr 30;382(18):1732-1738. doi: 10.1056/NEJMoa1917537. PMID 32348644
- [Background] Tan DW, Schiefer MA, Keith MW, Anderson JR, Tyler J, Tyler DJ. A neural interface provides long-term stable natural touch perception. Sci Transl Med. 2014 Oct 8;6(257):257ra138. doi: 10.1126/scitranslmed.3008669. PMID 25298320
- [Background] Schiefer MA, Graczyk EL, Sidik SM, Tan DW, Tyler DJ. Artificial tactile and proprioceptive feedback improves performance and confidence on object identification tasks. PLoS One. 2018 Dec 5;13(12):e0207659. doi: 10.1371/journal.pone.0207659. eCollection 2018. PMID 30517154
- [Background] Petrini FM, Valle G, Strauss I, Granata G, Di Iorio R, D'Anna E, Cvancara P, Mueller M, Carpaneto J, Clemente F, Controzzi M, Bisoni L, Carboni C, Barbaro M, Iodice F, Andreu D, Hiairrassary A, Divoux JL, Cipriani C, Guiraud D, Raffo L, Fernandez E, Stieglitz T, Raspopovic S, Rossini PM, Micera S. Six-Month Assessment of a Hand Prosthesis with Intraneural Tactile Feedback. Ann Neurol. 2019 Jan;85(1):137-154. doi: 10.1002/ana.25384. Epub 2018 Dec 24. PMID 30474259
- [Background] Raspopovic S, Capogrosso M, Petrini FM, Bonizzato M, Rigosa J, Di Pino G, Carpaneto J, Controzzi M, Boretius T, Fernandez E, Granata G, Oddo CM, Citi L, Ciancio AL, Cipriani C, Carrozza MC, Jensen W, Guglielmelli E, Stieglitz T, Rossini PM, Micera S. Restoring natural sensory feedback in real-time bidirectional hand prostheses. Sci Transl Med. 2014 Feb 5;6(222):222ra19. doi: 10.1126/scitranslmed.3006820. PMID 24500407
- [Background] Dietrich C, Nehrdich S, Seifert S, Blume KR, Miltner WHR, Hofmann GO, Weiss T. Leg Prosthesis With Somatosensory Feedback Reduces Phantom Limb Pain and Increases Functionality. Front Neurol. 2018 Apr 26;9:270. doi: 10.3389/fneur.2018.00270. eCollection 2018. PMID 29755399
- [Background] Naschitz JE, Lenger R. Why traumatic leg amputees are at increased risk for cardiovascular diseases. QJM. 2008 Apr;101(4):251-9. doi: 10.1093/qjmed/hcm131. Epub 2008 Feb 16. PMID 18281705
- [Background] Petrini FM, Bumbasirevic M, Valle G, Ilic V, Mijovic P, Cvancara P, Barberi F, Katic N, Bortolotti D, Andreu D, Lechler K, Lesic A, Mazic S, Mijovic B, Guiraud D, Stieglitz T, Alexandersson A, Micera S, Raspopovic S. Sensory feedback restoration in leg amputees improves walking speed, metabolic cost and phantom pain. Nat Med. 2019 Sep;25(9):1356-1363. doi: 10.1038/s41591-019-0567-3. Epub 2019 Sep 9. PMID 31501600
- [Background] Rathnayake A, Saboo A, Malabu UH, Falhammar H. Lower extremity amputations and long-term outcomes in diabetic foot ulcers: A systematic review. World J Diabetes. 2020 Sep 15;11(9):391-399. doi: 10.4239/wjd.v11.i9.391. PMID 32994867